CLINICAL TRIAL: NCT00402038
Title: A Double-Blind, Phase 3, Two-Week, Placebo Controlled Study of Methylnaltrexone(MNTX) for the Relief of Constipation Due to Opioid Therapy in Advance Medical Illness.
Brief Title: Study of Methylnaltrexone (MNTX) for the Relief of Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Tage Ramakrishna, MD, Progenics Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MNTX 302
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Advance Illness Patients With OIC

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: SC Methylnaltrexone
- Arm 2 (Placebo Comparator)
  Interventions: Drug: SC Placebo

INTERVENTIONS:
Drug: SC Methylnaltrexone — Dose 1
  Arms: Arm 1
Drug: SC Placebo
  Arms: Arm 2

SUMMARY:
To determine the efficacy of subcutaneous MNTX to relieve opioid-induced constipation in patients with advanced medical illness.

DETAILED DESCRIPTION:
This is a multi-center, double-blind, randomized parallel group study conducted in patients with advanced medical illness and opioid-induced constipation. Eligible patients are randomly assigned to receive SC doses of either MNTX, dose 1 or placebo every other day for 2 weeks. At Day 8, eligible patients, if allowed, could be escalated to a a higher dose of MNTX.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Negative pregnancy test (serum or urine) at screening for all women of childbearing potential
* Advanced Medical Illness (i.e., terminal illness, such as incurable cancer or end of stage AIDS) with life expectancy of ≥ 1 month
* patient must sign ICF

Exclusion Criteria:

* Women who are pregnant and/or nursing
* Previous treatment with MNTX
* Participation in any other studies involving investigational products within 30 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2004-02; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Laxation within four hours of a single dose of SC MNTX and efficacy of SC MNTX every other day over a 1 week period. | 2 weeks
  To determine the efficacy of a single dose of SC MNTX compared with placebo in inducing laxation within 4 hours.
  To determine the efficacy of SC MNTX every other day over a 1-week treatment period in relieving OIC in patients with AMI.

CONTACTS AND LOCATIONS:
Overall Officials: Tage Ramakrishna, MD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Inc., Tarrytown, New York, United States

REFERENCES:
- [Derived] Liao SS, Slatkin NE, Stambler N. The Influence of Age on Central Effects of Methylnaltrexone in Patients with Opioid-Induced Constipation. Drugs Aging. 2021 Jun;38(6):503-511. doi: 10.1007/s40266-021-00850-w. Epub 2021 Mar 31. PMID 33788162
- [Derived] Chamberlain BH, Rhiner M, Slatkin NE, Stambler N, Israel RJ. Subcutaneous methylnaltrexone for opioid-induced constipation in advanced-illness patients with or without active cancer. Pain Manag. 2020 Mar;10(2):73-84. doi: 10.2217/pmt-2019-0045. Epub 2020 Jan 17. PMID 31951150
- [Derived] Nalamachu SR, Pergolizzi J, Taylor R Jr, Slatkin NE, Barrett AC, Yu J, Bortey E, Paterson C, Forbes WP. Efficacy and Tolerability of Subcutaneous Methylnaltrexone in Patients with Advanced Illness and Opioid-Induced Constipation: A Responder Analysis of 2 Randomized, Placebo-Controlled Trials. Pain Pract. 2015 Jul;15(6):564-71. doi: 10.1111/papr.12218. Epub 2014 May 10. PMID 24815199
- [Derived] Lipman AG, Karver S, Cooney GA, Stambler N, Israel RJ. Methylnaltrexone for opioid-induced constipation in patients with advanced illness: a 3-month open-label treatment extension study. J Pain Palliat Care Pharmacother. 2011;25(2):136-45. doi: 10.3109/15360288.2011.573531. PMID 21657861
- [Derived] Thomas J, Karver S, Cooney GA, Chamberlain BH, Watt CK, Slatkin NE, Stambler N, Kremer AB, Israel RJ. Methylnaltrexone for opioid-induced constipation in advanced illness. N Engl J Med. 2008 May 29;358(22):2332-43. doi: 10.1056/NEJMoa0707377. PMID 18509120
- See also: Related Info — http://www.progenics.com